CLINICAL TRIAL: NCT05277207
Title: Tobacco Cessation Treatment Preferences Among Veteran Smokers (CDA 17-005)
Brief Title: Tobacco Cessation Treatment Preferences Among Veteran Smokers
Acronym: MESH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDX 22-005
Record Dates: First submitted 2022-03-02; First posted 2022-03-14 (Actual); Results first posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Tobacco Use
Keywords: tobacco use; smoking
MeSH Terms: conditions — Tobacco Use; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MESH (Experimental): Participants assigned to this group will receive a treatment that includes personalized smoking cessation facilitation meetings with cognitive-behavioral therapy, personalized smoking cessation pharmacotherapy, and personalized text messaging.
  Interventions: Behavioral: Personalized Smoking Cessation Facilitation Meetings; Drug: Personalized Smoking Cessation Pharmacotherapy; Behavioral: Personalized Text Messaging Support
- Best Practice Telehealth Group (Active Comparator): Participants assigned to this group will be referred to Quit Vet (VA's quitline for stopping tobacco) and SmokefreeVET (a free text messaging program to help you quit), and will receive information about getting quit medications.
  Interventions: Behavioral: SmokefreeVET; Behavioral: VA Quitline; Other: Education about pharmacotherapy

INTERVENTIONS:
Behavioral: Personalized Smoking Cessation Facilitation Meetings — Participants will participate in 5-7 meetings in which they will receive cognitive-behavioral therapy for tobacco cessation.
  Arms: MESH
Drug: Personalized Smoking Cessation Pharmacotherapy — Participants may receive pharmacotherapy for smoking cessation based on VA Pharmacy Benefits Management Services guidelines. Medications may include nicotine-replacement therapy, varenicline, and/or bupropion.
  Arms: MESH
Behavioral: Personalized Text Messaging Support — If the participant has a working cell phone and is willing to receive text messages, supportive, personalized text messages will be sent to the participant starting after Session 1 and extending through 6 months post-quit using VA's Annie texting capability.
  Other Names: Annie
  Arms: MESH
Behavioral: SmokefreeVET — Participants will receive a referral to SmokefreeVET, a text-messaging intervention designed to help veterans prepare for and attempt quitting smoking.
  Arms: Best Practice Telehealth Group
Behavioral: VA Quitline — Participants will receive a referral to VA Quitline, which is a nationally available telehealth intervention that provides assistance to veterans who wish to quit tobacco use. Quitline includes five sessions of cognitive-behavioral treatment.
  Arms: Best Practice Telehealth Group
Other: Education about pharmacotherapy — Participants will receive a handout that provides them with information about pharmacotherapies for tobacco cessation.
  Arms: Best Practice Telehealth Group

SUMMARY:
There are significant barriers to tobacco cessation treatment for patients and providers in specialty care clinical settings. Specialty providers cite several barriers to delivering evidence-based tobacco cessation care, including insufficient time and lack of training. In addition, a large proportion of patients who begin tobacco cessation treatment do not quit. Use of healthcare technology (i.e., telehealth, electronic health record, and computerized treatment algorithms based on patient data) to improve patients' ability to quit tobacco use. The purpose of this study is to demonstrate the feasibility of a larger trial, and to evaluate the acceptability of the intervention design. Thirty participants will be assigned to receive either 1) a treatment that includes personalized counseling, tobacco cessation medications, and text messaging; or 2) referral to Department of Veterans Affairs' Quitline program plus SmokefreeVET, a text messaging program.

DETAILED DESCRIPTION:
There are significant barriers to tobacco cessation treatment for patients and providers in specialty care clinical settings. Specialty providers in general cite several prominent barriers to delivering evidence-based tobacco cessation care, including insufficient time, lack of training, a perception of low motivation in their patients, and concerns about the sensitivity of tobacco cessation discussions. In addition, a large proportion of patients who begin tobacco cessation treatment do not achieve initial abstinence. Use of healthcare technology (i.e., telehealth, electronic health record, and computerized treatment algorithms based on patient data) to personalize treatment has the potential to increase patient engagement and proactively address treatment non-response. The proposed randomized controlled trial is a two-arm experimental design to demonstrate the feasibility of a larger trial and the acceptability of the intervention design. Participants (N = 30) will be stratified by clinic and randomized to either 1) the active treatment, which includes personalized cognitive behavioral treatment, personalized smoking cessation pharmacotherapy, and test messaging support; or 2) standard of care Department of Veterans Affairs' Quitline (telehealth intervention including 5 sessions of CBT) plus SmokefreeVET (text-messaging intervention).

ELIGIBILITY:
Inclusion Criteria:

* Durham VA patient
* willing to complete study procedures
* appointment in Durham VA Infectious Disease (ID) Clinic or Durham VA Cardiology Section within the past 12 months
* currently smoking 7 times per week (cigarettes, cigars, cigarillos, hookah, etc.) and/or using 1 can of smokeless tobacco per week

Exclusion Criteria:

* participation in Aim 3 (already received the intervention)
* current hospitalization (recent hospitalization is acceptable)
* currently not using combustible or smokeless tobacco (vaping only)
* acute risk for suicide documented in the medical record
* or inability to complete study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M. Wilson, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data sets will be available upon written FOIA request. Final data sets will also be maintained locally until enterprise-level resources become available for broader long-term storage and access unless the relevant ORD or VA Program Office Funding Announcement states otherwise.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MESH | Best Practice Telehealth Group
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MESH | Best Practice Telehealth Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (11.6) | 61.7 (10.2) | 59.75 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 14 | 14 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 9 | 19
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Report Post-treatment Satisfaction
Description: Post-treatment satisfaction will be measured at the 3-month follow-up. Satisfaction will be defined as a mean score greater than 3.5 on the satisfaction measure.
Time Frame: Post-treatment 3-month follow-up visit (approximately three months after enrollment)
Population: One control participant withdrew prior to the 3-month-follow-up, resulting in 14 control group participants.
Measure: Count of Participants; unit: Participants
Arm/Group | MESH | Best Practice Telehealth Group
Number analyzed (Participants) | 15 | 14
Participants | 15 | 10

2. Secondary Outcome: Treatment Attendance
Description: Treatment attendance is defined as the proportion of participants who complete at least one treatment session (via self-report for control group, via attendance logs for treatment group).
Time Frame: Post-treatment, approximately eight weeks after baseline visit
Measure: Count of Participants; unit: Participants
Arm/Group | MESH | Best Practice Telehealth Group
Number analyzed (Participants) | 15 | 14
Participants | 15 | 3

3. Secondary Outcome: Therapist-rated Treatment Acceptability in Active Treatment Group
Description: The proportion of post-treatment acceptability scores greater than 3.5 will be reported. Post-treatment therapist acceptability will be measured at the 3-month follow-up. Acceptability will be defined as a mean score greater than 3.5 on the acceptability measure.
Time Frame: Post-treatment 3-month follow-up visit (approximately three months after enrollment)
Population: Therapist-rated treatment acceptability was only measured in the active treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | MESH | Best Practice Telehealth Group
Number analyzed (Participants) | 15 | 0
Participants | 14 |

4. Secondary Outcome: Proportion of Participants Who Completed Treatment in the Active Treatment Group
Description: The investigators will provide the proportion of participants assigned to the active treatment group who complete treatment.
Time Frame: Post-treatment, approximately eight weeks after baseline visit
Population: This outcome was only measured in active treatment recipients
Measure: Number; unit: Percent pts completing treatment
Arm/Group | MESH | Best Practice Telehealth Group
Number analyzed (Participants) | 15 | 0
Percent pts completing treatment | 100 |

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | MESH | Best Practice Telehealth Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 3/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MESH (N=15) | Best Practice Telehealth Group (N=15)
Nausea due to nicotine replacement therapy (Gastrointestinal disorders) | 1 (1) | 0 (0)
mood symptoms related to Varenicline use (Psychiatric disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT05277207/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT05277207/ICF_000.pdf